CLINICAL TRIAL: NCT05725915
Title: Multiparameter Prediction Model of Immune Checkpoint Inhibitors Combined With Chemotherapy in Advanced Non-small Cell Lung Cancer: a Real-world Study
Brief Title: Prediction Model of ICIs Combined With Chemotherapy in Advanced NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Red Clove Public Welfare Development Center (Other)
Responsible Party: Sponsor
Other Study IDs: BJ-HDX-20220781
Record Dates: First submitted 2023-01-16; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer, Nonsmall Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The reliable predictive markers to identify which patients with advanced non-small cell lung cancer tumors will achieve durable clinical benefit for chemo-immunotherapy are needed. This study is a real world study, aiming to establish a multi-parameter model to predict the efficacy of immune checkpoint inhibitor(ICI) combined with chemotherapy, and to explore the correlation and predictive value of each single biomarker, so as to assist physician to select patients who may benefit for a long time as early as possible and guide clinical accurate treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female, ≥18 years old;
2. Patients with a definite cytological or histopathological diagnosis of non-small cell lung cancer;
3. Locally advanced (stage IIIB/IIIC) or metastatic (stage IV) NSCLC unable to receive radical surgery and/or radical radiotherapy (with or without concurrent chemotherapy) (AJCC cancer stage 8 clinical stage)
4. There is no known ALK gene translocation
5. For patients with EGFR-negative non-squamous cell carcinoma, or patients with EGFR-negative/unknown squamous cell carcinoma, it is required that they have not received systemic antitumor therapy for advanced NSCLC in the past (patients have received neoadjuvant chemotherapy, adjuvant chemotherapy, radiotherapy or chemoradiotherapy for curing non-metastatic disease in the past, A disease-free interval of ≥6 months was required between the last chemotherapy and/or radiotherapy).
6. Patients with non-squamous cell carcinoma with EGFR-sensitive mutation and EGFR TKI progression could be enrolled if they met any of the following requirements:

   Progress in Treatment of 1/2 generation EGFR TKI, T790M-; EGFR TKI treatment progress of 1/2 generation, T790M+, after 3 generations of EGFR TKI treatment progress again; T790M status was not considered in patients who had progressed to the initial 3 generations of EGFR TKI therapy.
7. At least 1 measurable lesion according to RECIST 1.1
8. Receiving immune checkpoint inhibitor therapy for more than 2 cycles
9. ECOG PS 0-1 score
10. Be able to understand and abide by the requirements of the agreement, and voluntarily participate in the study.

Exclusion Criteria:

1. Patients participating in other clinical studies;
2. Patients with serious lack of diagnosis and treatment data;
3. Patients could not understand the purpose of the study or disagreed with the requirements of the study;
4. A history of other tumors within 5 years;
5. Patients judged by the researchers as not suitable for inclusion in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with inoperable stage IIIB to IV NSCLS using immune checkpoint inhibitors in combination with chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival（PFS）in days | From date of enrollment until the date of first documented progression, assessed up to 2 years.
  the time between the time a patient with tumor disease begins treatment and the time when disease progression is observed or death from any cause occurs.

SECONDARY OUTCOMES:
ctDNA in concentration | The First treatment (month 1), the second treatment (month 2) and the time of progression (assessed up to 2 years)
  The best predictive value of ctDNA concentration change threshold and the best collection time.

CONTACTS AND LOCATIONS:
Overall Officials: Shuhua Han, docter, Study Chair — Southeast University Zhongda Hospital
Locations (1):
- Shuhua Han, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
This is the initial stage of the study, and the data sets generated and analyzed in the later stage of the study can be obtained from corresponding authors according to reasonable requirements.